CLINICAL TRIAL: NCT01213953
Title: Isolation and Authentication of Mesenchymal Stem Cell-like Progenitor Cells From the Degenerated Intervertebral Disc of Lumbar Spine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsieh-Hsing Lee, Department of Orthopedics, Shuang Ho Hospital, Taipei Medical University
Other Study IDs: 98025
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Lower Back Pain; Disc Degeneration
Keywords: Vertebral disc, mesenchymal stem cell.
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biospecimen is the tissue waste after the surgery of discectomy.
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed for evaluating the presence of mesenchymal stem cells of vertebral disc. Isolation and authentication of these cells may be applied for the vertebral disc regeneration and the research tissue engineering.

DETAILED DESCRIPTION:
We will collect the degenerative disc from adults and isolate the mesenchymal stem cell-like precursors cells. The function of osteogenic, chondrogenic, and lipogenic differentiation will be authenticated. The results will offer the information for cell source of tissue engineering in the future.

ELIGIBILITY:
Inclusion Criteria:

* The adults with disc degeneration（age >= 20 years old） A. Herniated intervertebral disc. B. Spondylolisthesis. C. Spondylolysis. D. Other causes of disc degeneration.

Exclusion Criteria:

* Age < 20 years old.
* Pregnancy.
* Spinal tumors.
* Spinal infections.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients received the surgery of discectomy for the degenerative disc.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh-Hsing Lee, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan